CLINICAL TRIAL: NCT05451719
Title: Efficacy and Safety of Fruquintinib Plus Capecitabine Versus Capecitabine as Maintenance Treatment for Metastatic Colorectal Cancer After First-line Chemotherapy: A Phase II, Randomized, Controlled Study
Brief Title: Fruquintinib Plus Capecitabine Versus Capecitabine as Maintenance Therapy for Metastatic Colorectal Cancer After First-line Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junjie Peng, Chief Physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C116
Record Dates: First submitted 2022-07-02; First posted 2022-07-11 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer; Colorectal Cancer Stage IV
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fruquintinib Plus Capecitabine (Experimental): Maintenance therapy with Fruquintinib Plus Capecitabine
  Interventions: Drug: Fruquintinib Plus Capecitabine
- Capecitabine (Active Comparator): Maintenance therapy with Capecitabine
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Fruquintinib Plus Capecitabine — Fruquintinib at the dose determined in phase safety lead-in, orally once daily, on d1-21, given every 4 weeks (Q4W). Capecitabine at the dose 850mg/m2, orally twice daily, d1-7 and d15-21, given every 4 weeks (Q4W)
  Arms: Fruquintinib Plus Capecitabine
Drug: Capecitabine — Capecitabine at the dose 850mg/m2, orally twice daily, d1-7 and d15-21, given every 4 weeks (Q4W)
  Arms: Capecitabine

SUMMARY:
This is an open-label, multicenter, randomized phase 2 study evaluating the efficacy and safety of fruquintinib plus capecitabine versus capecitabine as maintenance therapy for metastatic colorectal cancer after first-line treatment. Patients who have already achieved disease control (including CR/PR and SD) after ≥6 cycles of standard first-line induction treatment, and are still unresectable would be assigned into 2 maintenance treatment groups by randomization in a 1:1 ratio to receive fruquintinib + capecitabine or capecitabine. All patients will be treated until progressive disease, death from any cause, unacceptable toxicity or informed consent withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old at the time of signing the informed consent;
2. Patients who have been histologically or cytologically confirmed adenocarcinoma of the colon or rectum (stage IV);
3. Patients who have achieved disease control (including CR/PR and SD) after 6 cycles of first-line standard chemotherapy and are still unresectable;
4. At least one measurable metastatic lesion(s) as defined by RECIST version 1.1;
5. ECOG performance status of 0-2;
6. Life expectancy≥3 months;
7. Adequate organ and bone marrow functions: Neutrophils >1.5×109/L, platelets >100×109/L, and hemoglobin >9 g/dL; Total bilirubin <1.5×upper limit of normal (ULN); aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and/or alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) <3×ULN (<5×ULN in case of liver metastases); Creatinine clearance (calculated according to Cockcroft and Gault) ≥60 mL/min; Serum creatinine < 1.5×ULN;
8. Women of childbearing age must have a negative pregnancy test within the first day of the study, and contraceptive methods should be taken during the study until 6 months after the last administration;
9. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

1. Had a surgical procedure within 4 weeks prior to treatment; Received radiation therapy, radiofrequency therapy, chemotherapy, immunotherapy or molecular targeted therapy, or other investigational drugs within 2 weeks prior to treatment;
2. Prior treatment with anti-vascular small-molecule targeted drugs, such as Fruquintinib or Regorafenib;
3. A history of severe intolerance to capecitabine or 5-FU (i.e. grade 4 toxicity of one of the drugs; Grade 3-4 toxicity of other concomitant drugs is not excluded);
4. Symptomatic brain or meningeal metastases (except for patients with BMS who have received local radiotherapy or surgery for more than 6 months and whose disease is stable).
5. Patients with hypertension that cannot be well controlled by antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
6. Have obvious clinical bleeding symptoms or obvious bleeding tendency within 3 months before treatment (bleeding > 30 mL within 3 months, hematemesis, black feces, hematozoia), hemoptysis (fresh blood > 5 mL within 4 weeks), etc. Treatment for venous/venous thrombosis events within the previous 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; Long-term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day);
7. Active heart disease, including myocardial infarction, severe/unstable angina, 6 months prior to treatment. Echocardiography examination left ventricular ejection fraction < 50%, arrhythmia control is not good;
8. The patient has had other malignant tumors within 3 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
9. Allergy to the study drug or any of its excipients;
10. Severe infection with active or uncontrolled infection;
11. Any other disease, with clinical significance of metabolic abnormalities, abnormal physical examination or laboratory abnormalities, according to researchers, there is reason to suspect the patient has not suitable for the use of study drugs of a disease or condition (such as have a seizure and require treatment), or will affect the interpretation of results, or to make patients in high-risk situations;
12. Urine routine showed urine protein ≥2+, and 24-hour urine protein level >1.0g.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | From Baseline to primary completion date, about 24 months
  A duration from the date of initial treatment to disease progression or death of any cause

SECONDARY OUTCOMES:
Objective response rate (ORR, RECIST 1.1) | From Baseline to primary completion date, about 24 months
  The incidence of confirmed complete response or partial response
Disease Control Rate (DCR, RECIST 1.1) | From Baseline to primary completion date, about 24 months
  The incidence of complete response, partial response and stable disease
Overall survival (OS) | From Baseline to primary completion date, about 24 months
  From the time of enrollment to death caused by any reason
The incidence of adverse events | From Baseline to primary completion date, about 24 months
  The safety and tolerability of Surufatinib will be evaluated based on adverse events data.

IPD SHARING:
Plan to Share IPD: No